CLINICAL TRIAL: NCT04101747
Title: To Explore the Diversity of Intestinal Flora in Patients With Advanced Hepatocellular Carcinoma Receiving Anti-PD-1 Combined With Targeted Drug Therapy and the Correlation Between Metabolites and Therapeutic Effect:A Multi-Center Study
Brief Title: To Explore the Diversity of Intestinal Flora in Patients With Advanced HCC Combin ed With Anti-PD-1 and Targeted Drug Therapy and the Correlation Between Metabolites and Therapeutic Effect
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, Professor of department of infectious disease Third Affiliated Hospital,Sun Yat-Sen University, Sun Yat-sen University
Other Study IDs: XC2
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced hepatocellular carcinoma; Combination of PD-1/PD-L1 Inhibitors and Targeted Drugs; Diversity of intestinal flora; Metabolites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before the treatment of PD-1 (no more than 24 hours), during the treatment of PD-1 (every time before treatment, three weeks treatment, a total of 11 follow-up visits), at the end of treatment, fecal samples were collected in sterile containers for 5-10 g, feces were stored at 4 C, frozen at - 80 C within 24 hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is to explore the correlation between intestinal flora diversity and meta bolites in patients with advanced lver cancer rceiving Anti-PD-1 combined target-ed drug therapy,so that to get the analysis of intestinal flora of PD-1 inhibitors in liver cancer.

DETAILED DESCRIPTION:
The combination of PD-1/PD-L1 inhibitors and targeted drugs as a promising strategy for the treatment of hepatocellular carcinoma has a breakthrough significance for the treatment of some advanced and refractory tumors.However,studies have shown that intestinal flora diversity indicates a good prognosis of PD-1/PD-L1 inhibitors in the treatment of non-small cell lung cancer, the intestinal flora analysis of PD-1 inhibitors in hepatocellular carcinoma is still a new field to be explored.

This study is to select patients who meet the criteria of entry and discharge, sign informed consent, obtain patients'clinical data, pathological and case data, and enter the database. Before the treatment of PD-1 (no more than 24 hours), during the treatment of PD-1 (every time before treatment, three weeks, a total of 11 follow-up visits), at the end of treatment, fecal samples were collected in sterile containers for 5-10g, and feces were stored at 4 degrees C, frozen at - 80 degrees C within 24 hours; the response to treatment was evaluated every 6 weeks, and the disease was first evaluated clinically. The patients were divided into response group (R) (partial response or stable condition) or non-response group (NR) (disease progression) according to RECIST 1.1 evaluation criteria. Subgroup had high diversity of bacteria and low diversity of bacteria, and were observed continuously until the end of treatment. The bacterial ribosomal DNA was extracted, metabolites were detected and flow cytometry was used to analyze the data. The baseline intestinal microflora diversity, microflora diversity mapping, continuous Shannon index curve change mapping were compared between groups and within groups, and correlation validation was carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients signed informed voluntary enrollment and expected survival of more than 12 weeks;
* Patients with HCC confirmed by histopathology or cytology or clinic are HBV-related HCC;
* No systematic treatment for HCC has been received in the past, excluding local chemotherapy drugs used in TACE/TAI;
* Not suitable for surgical treatment;
* Child-Pugh Class: Grade A or B (≤7 points);
* BCLC stage C;
* ECOG PS≤1;
* At least one measurable lesion (according to RECIST v1.1 requirement, the length of spiral CT of the lesion is ≥10mm or the short diameter of enlarged lymph nodes is ≥15 mm);
* Organ Function Requirements (within 7 days before treatment):

Blood routine examination: WBC (>1.5 *109/L); PLT (>75 *109/L); HB (>90 g/L); no blood transfusion within 14 days before screening, G-CSF drug correction) Liver function tests: ALB (> 29 g/L); TBiL (< 1.5 * ULN); ALT, AST, AKP (< 5 * ULN); INR (< 2.3) or PT (< 6 seconds) exceeding normal control Renal function: Cr < 1.5 ULN or CCr > 50 mL/min

* Patients with active hepatitis B virus (HBV) infection: must receive anti HBV treatment;
* Fertility women should abstinence or use reliable methods of contraception during the observation of curative effect. Serum HCG test must be negative within 7 days before the study treatment, and must be non-lactating. When it comes to abstinence, partners should also have reliable and effective contraception;
* Assessment of patients who are eligible for anti-PD-1 combined with targeted drug therapy;
* Consent to sign informed consent and follow up for a long time.

Exclusion Criteria:

* Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously;
* Patients with moderate or severe ascites need therapeutic puncture and drainage or Child score > 2 (except those with small amount of ascites without clinical symptoms);
* Patients with a history of gastrointestinal bleeding or risk of bleeding within 6 months before the start of the study, such as severe esophageal varices, locally active gastrointestinal ulcer lesions, and positive persistent fecal occult blood;
* Known hereditary or acquired bleeding or thrombotic tendency, thrombosis or embolism occurred within 6 months before treatment, and aspirin > 325 mg/day was taken within 10 days before treatment;
* It is known that there is a history of severe allergy to any monoclonal antibody or anti-angiogenesis targeted drug;
* Severe infections occurred within 4 weeks before the start of the study, including but not limited to hospitalization due to infections, bacteremia or complications of severe pneumonia;
* Previous treatment with other anti-PD-1 antibodies or other immunotherapy against PD-1/PD-L1;
* Complicated with other hepatitis virus infection or alcoholic liver disease, hereditary metabolic liver disease, autoimmune liver disease and other liver diseases;
* Congenital or acquired immunodeficiency (HIV, or treatment with immunosuppressive agents or systemic hormones within 14 days before treatment (>10mg/d prednisone or other hormones)
* There are cardiopulmonary diseases that can not be well controlled, such as cardiac insufficiency above NYHA II or LVEF < 50% by color Doppler echocardiography, COPD with repeated pulmonary infections.
* Intravenous antibiotics or prophylactic antibiotics were given in the past month. -Receive immunopotentiation therapy, such as thymosin, Ridaxian, etc.
* Other factors that may affect the results of the study or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring combined treatment, accompanied by family or social factors, may affect patient safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Include patients who meet the entry and discharge criteria, obtain patients'clinical data, pathological and case data, enter the database, collect fecal samples of 5-10g, evaluate the response to treatment every 6 weeks, and conduct data analysis, compare the baseline intestinal microflora diversity between and within groups, microflora diversity mapping, continuous Shannon fingers. Number curve mapping, attention to follow-up patients, record treatment, progress, other toxic and side effects and combined drug use information.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (RR) | Up to approximately 3 years
  To analyse the Objective response rate (RR) of patients with advanced HCC receiving anti-PD-1 combined with targeted drug therapy
Disease control rate (DCR) | Up to approximately 3 years
  To exprole the Disease control rate (DCR) of patients with advanced HCC receiving anti-PD-1 combined with targeted drug therapy
Number of intestinal flora | Up to approximately 3 years
  To exprole the Number of intestinal flora of patients with advanced HCC receiving anti-PD-1 combined with targeted drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Chan Xie, Professor, Principal Investigator — The Third Affliated Hosoital of Sun Yat-Sun University